CLINICAL TRIAL: NCT04128358
Title: Triple Therapy in Patients With Idiopathic Thrombocytopenic Purpura : What is Behind?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Safaa AA Khaled, Clinical Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Skhaled21
Record Dates: First submitted 2019-10-13; First posted 2019-10-16 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Idiopathic Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Intervention Model Description: This is a randomized clinical trial aimed to assess the effect of strong immunosuppression in patients with ITP on Triple therapy on acquiring viral hepatitis infection C or B.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group on high dose dexamethasone, cyclosporin and rituximab (Experimental): Egyptian patients with idiopathic thrombocytopenic purpura on high dose dexamethasone together with cyclosporine and rituximab.
  Interventions: Diagnostic Test: Serological assay for blood born viral hepatitis; Diagnostic Test: Quantitative microbiological test for HCV
- Group on steroids only (Active Comparator): Egyptian patients with idiopathic thrombocytopenic purpura on parenteral or oral steroids.
  Interventions: Diagnostic Test: Serological assay for blood born viral hepatitis; Diagnostic Test: Quantitative microbiological test for HCV
- Placebo group (Placebo Comparator): Egyptian normal healthy volunteers who share on the President Initiative (100 Million Health).
  Interventions: Diagnostic Test: Serological assay for blood born viral hepatitis; Diagnostic Test: Quantitative microbiological test for HCV

INTERVENTIONS:
Diagnostic Test: Serological assay for blood born viral hepatitis — Qualitative PCR for patients with hepatitis C antibody positive
  Other Names: Qualitative Polymerase chain reaction (PCR)
Diagnostic Test: Quantitative microbiological test for HCV — Quantitative PCR in those with proven HCV infection

SUMMARY:
Idiopathic thrombocytopenic purpura (ITP) is a benign hematological disorder characterized by isolated thrombocytopenia. Development of antiplatelet autoantibodies is the main pathogenetic mechanism in patients with ITP. However the exact pathogenesis of ITP is complex in which megakaryocyte immune injury and T-cell mediated platelet destruction play significant role. Accordingly treatment of ITP relies mainly on immunosuppression. Recently triple regimen of high dose dexamethasone together with cyclosporine and rituximab was found to induce prolonged remission in patients with ITP compared with single agent immunosuppression. On the other hand this regimen suppresses all immune cells thus predisposing patient to serious infections, which is the main cause of morbidity in ITP furthermore infection enhances autoimmunity.

This study will focus on viral hepatitis C and B infection in Egyptian patients with idiopathic thrombocytopenic purpura on Triple therapy and aims to:

* Assess and improve preventive measures of blood born hepatitis infection in the hematology ward in Egypt.
* Investigate influence of immunosuppression on infection with blood born hepatitis on Egyptian patients with ITP on Triple therapy.
* Study the impact of blood born hepatitis infection on clinical outcome on those patients.
* Identify risk factors and routes of transmission of blood born viral hepatitis in the hematology ward in Egypt

DETAILED DESCRIPTION:
Blood born viral hepatitis is a type of viral hepatitis that is usually transmitted with transfusion of blood and blood products. Accordingly patients with hematological disorders are at higher risk for infection with blood born hepatitis as blood transfusion besides regular sampling are integral parts in management of hematological patients. This was the case in patients with ITP, however not all patients with ITP in need for regular platelet transfusion. The mainstay of treatment of ITP is immunosuppression, that was mainly dependent on parenteral or oral steroids for long time. Triple therapy was recently introduced for treatment of patients with ITP it induces strong immunosuppression that could make patients vulnerable to infections.

Several studies accused immunosuppression in patients with hematological malignancies under chemotherapy to be a risk factor for infection with blood born hepatitis, as such triple therapy could predispose patients with ITP to blood born viral hepatitis infection.

On the other hand infection with blood born hepatitis in patients with ITP on Triple therapy could affect patient outcome and response to treatment. This is because thrombocytopenia is a common extra hepatic manifestation of hepatitis C viral infection on its chronic form.

Egypt is a country with high prevalence of blood born viral hepatitis viral hepatitis C. Recently, the president of Egypt elaborated an initiative (100 million Health) that was managed with the Ministry of Health in all over the country. This initiative aimed to eliminate blood born hepatitis particularly C from the Country.

This work will be conducted in Egypt and focused on ITP patients on Triple therapy to assess their vulnerability for infection with blood born hepatitis as they are a particular sector of the Egyptian population at higher risk for infection.

ELIGIBILITY:
Inclusion Criteria:

* Normal healthy Egyptians on the age range from 18-85.
* Egyptian patients with ITP in age range from 18- 65 on high dose dexamethasone together with cyclosporin and rituximab .
* Egyptian patients with ITP in age range from 18- 65 on parenteral or oral steriods.

Exclusion Criteria:

* Age less than 18 years old.
* Pregnancy
* Thrombocytopenia other than ITP.
* Patients with ITP but on other modalities of treatment.
* Patients with blood born viral hepatitis infection before treatment with high dose dexamethasone together with cyclosporin and rituximab

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Incidence | 6-months
  Number of ITP patients on Triple therapy became infected with blood born viral hepatitis.
Platelet count | 6-months
  Number of ITP patients on Triple therapy infected with HCV or HBV and their platelet count
Primary prevention | One month
  Number of medical and paramedical staff who follow preventive measures for HCV and HBV in the hematology ward before and after an educational program
Risk factors | 6-months
  Number of ITP patients who became infected with HCV or HBV after exposure to a risk factor

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed El yamany, Prof., Study Director — Assiut University; Shymaa M Nageeb, MD, Principal Investigator — Assiut University; Eman NaserEldin, Prof, Principal Investigator — Assiut University; Ahmed Khair, Ass. Prof., Study Director — faculty of medicine
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodeghiero F, Stasi R, Gernsheimer T, Michel M, Provan D, Arnold DM, Bussel JB, Cines DB, Chong BH, Cooper N, Godeau B, Lechner K, Mazzucconi MG, McMillan R, Sanz MA, Imbach P, Blanchette V, Kuhne T, Ruggeri M, George JN. Standardization of terminology, definitions and outcome criteria in immune thrombocytopenic purpura of adults and children: report from an international working group. Blood. 2009 Mar 12;113(11):2386-93. doi: 10.1182/blood-2008-07-162503. Epub 2008 Nov 12. PMID 19005182
- [Background] Kuwana M, Ikeda Y. The role of autoreactive T-cells in the pathogenesis of idiopathic thrombocytopenic purpura. Int J Hematol. 2005 Feb;81(2):106-12. doi: 10.1532/ijh97.04176. PMID 15765777
- [Background] Patel VL, Mahevas M, Lee SY, Stasi R, Cunningham-Rundles S, Godeau B, Kanter J, Neufeld E, Taube T, Ramenghi U, Shenoy S, Ward MJ, Mihatov N, Patel VL, Bierling P, Lesser M, Cooper N, Bussel JB. Outcomes 5 years after response to rituximab therapy in children and adults with immune thrombocytopenia. Blood. 2012 Jun 21;119(25):5989-95. doi: 10.1182/blood-2011-11-393975. Epub 2012 May 7. PMID 22566601
- [Background] Gudbrandsdottir S, Birgens HS, Frederiksen H, Jensen BA, Jensen MK, Kjeldsen L, Klausen TW, Larsen H, Mourits-Andersen HT, Nielsen CH, Nielsen OJ, Plesner T, Pulczynski S, Rasmussen IH, Ronnov-Jessen D, Hasselbalch HC. Rituximab and dexamethasone vs dexamethasone monotherapy in newly diagnosed patients with primary immune thrombocytopenia. Blood. 2013 Mar 14;121(11):1976-81. doi: 10.1182/blood-2012-09-455691. Epub 2013 Jan 4. PMID 23293082
- [Background] Polaris Observatory HCV Collaborators. Global prevalence and genotype distribution of hepatitis C virus infection in 2015: a modelling study. Lancet Gastroenterol Hepatol. 2017 Mar;2(3):161-176. doi: 10.1016/S2468-1253(16)30181-9. Epub 2016 Dec 16. PMID 28404132
- [Background] Kouyoumjian SP, Chemaitelly H, Abu-Raddad LJ. Characterizing hepatitis C virus epidemiology in Egypt: systematic reviews, meta-analyses, and meta-regressions. Sci Rep. 2018 Jan 26;8(1):1661. doi: 10.1038/s41598-017-17936-4. PMID 29374178
- [Background] Wedemeyer H, Duberg AS, Buti M, Rosenberg WM, Frankova S, Esmat G, Ormeci N, Van Vlierberghe H, Gschwantler M, Akarca U, Aleman S, Balik I, Berg T, Bihl F, Bilodeau M, Blasco AJ, Brandao Mello CE, Bruggmann P, Calinas F, Calleja JL, Cheinquer H, Christensen PB, Clausen M, Coelho HS, Cornberg M, Cramp ME, Dore GJ, Doss W, El-Sayed MH, Ergor G, Estes C, Falconer K, Felix J, Ferraz ML, Ferreira PR, Garcia-Samaniego J, Gerstoft J, Giria JA, Goncales FL Jr, Guimaraes Pessoa M, Hezode C, Hindman SJ, Hofer H, Husa P, Idilman R, Kaberg M, Kaita KD, Kautz A, Kaymakoglu S, Krajden M, Krarup H, Laleman W, Lavanchy D, Lazaro P, Marinho RT, Marotta P, Mauss S, Mendes Correa MC, Moreno C, Mullhaupt B, Myers RP, Nemecek V, Ovrehus AL, Parkes J, Peltekian KM, Ramji A, Razavi H, Reis N, Roberts SK, Roudot-Thoraval F, Ryder SD, Sarmento-Castro R, Sarrazin C, Semela D, Sherman M, Shiha GE, Sperl J, Starkel P, Stauber RE, Thompson AJ, Urbanek P, Van Damme P, van Thiel I, Vandijck D, Vogel W, Waked I, Weis N, Wiegand J, Yosry A, Zekry A, Negro F, Sievert W, Gower E. Strategies to manage hepatitis C virus (HCV) disease burden. J Viral Hepat. 2014 May;21 Suppl 1:60-89. doi: 10.1111/jvh.12249. PMID 24713006
- [Background] Wang CS, Yao WJ, Wang ST, Chang TT, Chou P. Strong association of hepatitis C virus (HCV) infection and thrombocytopenia: implications from a survey of a community with hyperendemic HCV infection. Clin Infect Dis. 2004 Sep 15;39(6):790-6. doi: 10.1086/423384. Epub 2004 Aug 27. PMID 15472809
- [Background] Aref S, Sleem T, El Menshawy N, Ebrahiem L, Abdella D, Fouda M, Samara NA, Menessy A, Abdel-Ghaffar H, Bassam A, Abdel Wahaab M. Antiplatelet antibodies contribute to thrombocytopenia associated with chronic hepatitis C virus infection. Hematology. 2009 Oct;14(5):277-81. doi: 10.1179/102453309X439818. PMID 19843383
- [Background] Ennishi D, Terui Y, Yokoyama M, Mishima Y, Takahashi S, Takeuchi K, Okamoto H, Tanimoto M, Hatake K. Monitoring serum hepatitis C virus (HCV) RNA in patients with HCV-infected CD20-positive B-cell lymphoma undergoing rituximab combination chemotherapy. Am J Hematol. 2008 Jan;83(1):59-62. doi: 10.1002/ajh.21022. PMID 17712791